CLINICAL TRIAL: NCT04143750
Title: The Mass Balance and Biotransformation Study of [14C] Vicagrel in Chinese Healthy Adult Male Volunteers
Brief Title: The Mass Balance and Biotransformation of [14C] Vicagrel in Healthy Man
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-MB-WKGL-08
Record Dates: First submitted 2019-10-21; First posted 2019-10-29 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Healthy Male Adult

STUDY DESIGN:
Intervention Model Description: single arm with single dose of 20mg vicagrel, containing about 120μCi [14C]Vicagrel
Masking Description: unrandomization and open labeled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]Vicagrel (Experimental)
  Interventions: Drug: [14C]Vicagrel

INTERVENTIONS:
Drug: [14C]Vicagrel — Take a suspension of 20 mg vicagrel ,containing about 120 μCi [14C]Vicagrel, in fasting within 5 minutes

SUMMARY:
This study was designed to evaluate the mass balance and biotransformation after single-dose of [14C]Vicagrel orally in Chinese healthy male volunteers, revealing the overall pharmacokinetic characteristics of vicagrel in humans, and providing a reference for the rational administration.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male adult.
* Age is between 18 and 45, inclusive.
* Body mass index is between 19 and 26, inclusive.
* Voluntarily to provide informed consent form.
* Willing and able to communicate with investigators and complete the trial according to clinical trial protocol.

Exclusion Criteria:

* Any abnormal and clinical significant findings to physic exam, vital sign, electrocardiogram, X-ray exam for chest, laboratory exam including blood biochemical, blood routine, blood coagulation, urine routine, routine stool plus occult blood and thyroid stimulating hormone, and so on.
* A positive examination result of HBsAg/HBeAg, HIV antibody and treponema pallidum antibody.
* Volunteers who take any medicines including OTC, hormone birth control and/or alternative medicines such as medicated diets, Chinese herbal medicines, hemostatics or supplements within 14 days before the screening.
* Volunteers have clinical product administration or clinical trial participation within 3 months before the screening.
* Any history of clinical serious disease, or presence illness/condition that, in the opinion of the investigator, would jeopardize the study results, including but not limited to the circulatory system, endocrine system, nervous system, digestive system, urinary system or history of blood, immune, mental and metabolic diseases.
* History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsade ventricular tachycardia, ventricular tachycardia, QT prolongation syndrome, or QT prolongation Symptoms and family history ,indicated by genetic evidence or sudden death of a close relative due to cardiac conditions at a young age.
* Volunteers or their immediate family have coagulopathy, coagulative/hemorrhagic disease ,such as hemophilia, gastrointestinal bleeding, cyanosis, coagulative /hemorrhagic symptoms ,such as hematemesis, melena, severe or recurrent epistaxis, hemoptysis, obvious hematuria or intracranial hemorrhage, coagulative/hemorrhagic family history, suspected vascular malformations, such as aneurysm or early onset stroke, CVA < 65 years old, bleeding tendency ,such as repeated bleeding gums, or previous active pathological bleeding.
* Current or recent (<6 months) disease of dyspepsia, esophageal reflux, stomach bleeding, peptic ulcer, often heartburn over one times every week or any surgery that may affect drug absorption , such as cholecystectomy.
* Major surgery or surgical incision did not completely heal within 6 months before the screening. Major surgery includes, but is not limited to, any volunteer with significant bleeding risk, prolonged general anesthesia, incision of a biopsy or significant traumatic injury.
* Ecchymoses were detected in the skin during physical examination.
* The prothrombin time (PT) and/or activated partial thromboplastin time (APTT) exceeds the upper limit of the normal range, or the hematocrit (HCT) or platelet count (PLT) is out of the normal range.
* Volunteers who are allergic to drugs, the same type of investigational product ,such as clopidogrel, ticagrelor, etc., pharmaceutical excipients, alcohol, food ingredients. Or who has special requirements for diet and cannot comply with the required diet.
* Suffering acne or perianal disease in blood in the stool or regularly.
* Volunteers have habitual constipation, diarrhea, irritable bowel syndrome or inflammatory bowel disease.
* Volunteers are alcoholism, often drinking in six months before screening which means more than 14 units of alcohol every week, or the alcohol breath test result is positive in screening. One unit alcohol equals 360 mL of beer, 45 mL of 40% alcohol or 150 mL of wine.
* Volunteers have daily smoking exceeds 5 cigarettes in three months before screening, or habitual use of nicotine products, and can not be withdrawn during the trial.
* Abusing drug, using soft drugs such as marijuana three months prior to screening, using hard drugs such as cocaine, amphetamine, phencyclidine, etc. one year prior to screening; or urine test for drugs is positive in screeing.
* Volunteers have habitual drinking of grapefruit juice, excessive tea, coffee and/or caffeinated beverages, and who can not be abstained during the trial.
* Volunteers who have to work in radioactive conditions in long time, participated in radio-labeled drug clinical trial or had significant radioactive exposure within one year before the trial, more than 2 times of chest/abdominal CT, or more than 3 times of different types of X-ray exam.
* Volunteer and their spouse who have a birth plan or who are unwilling to take strict contraceptive measures such as condoms, contraceptive sponges, contraceptive gels, contraceptive film, intrauterine device, contraceptive for oral and injection, subcutaneous implant, etc., during the trial or in the future one year after the trial.
* Volunteers, who have had blood loss/donation up to 400 mL within 3 months before the screening, or received blood transfusion within 1 month.
* Volunteers are not suitable for this clinical trial, in the opinions of investigators.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Total radioactive datas in blood | from 0 hour to 240 hours after administration
  Total radioactive distribution and pharmacokinetics in blood and plasma
Total radioactive datas in excreta | from 0 hour to 240 hours after administration
  Total radioactive distribution and pharmacokinetics in urine and feces; the main routes of [14C]Vicagrel excretion in human
Peak Plasma Concentration (Cmax) | from 0 hour to 240 hours after administration
  Determine the Cmax of Vicagrel metabolites M3, M9-2, M15-1 and M15-2 in plasma
Area under the plasma concentration versus time curve (AUC) | from 0 hour to 240 hours after administration
  Determine the AUC of Vicagrel metabolites M3, M9-2, M15-1 and M15-2 in plasma
Time of Peak Plasma Concentration(Tmax) | from 0 hour to 240 hours after administration
  Determine the Tmax of Vicagrel metabolites M3, M9-2, M15-1 and M15-2 in plasma
Drug half-life in plasma(t1/2) | from 0 hour to 240 hours after administration
  Determine the T1/2 of Vicagrel metabolites M3, M9-2, M15-1 and M15-2 in plasma
Mean Residence Time (MRT) | from 0 hour to 240 hours after administration
  Determine the MRT of Vicagrel metabolites M3, M9-2, M15-1 and M15-2 in plasma
Numbers of Vicagrel Metabolites | from 0 hour to 240 hours after administration
  Detect Vicagrel Metabolites in blood, feces and urines as much as possible to clear the main routes of biotransformation

SECONDARY OUTCOMES:
Adverse Events | through the completion of study, an average of 2 months
  Review the relationship between investigational products and all the abnormal and clinically significant findings

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, PhD, Principal Investigator — First Affiliated Hospital of Suzhou Medical College
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China